CLINICAL TRIAL: NCT02694913
Title: Polymorphisms at Distinct Genetic Loci Affect Response to Anti-CD20 Monoclonal Antibody Therapies
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 1503016060
Record Dates: First submitted 2016-02-23; First posted 2016-03-01 (Estimated); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood will be taken to measure B-cell depletion. Any remaining sample will be stored for 15 years in the biobank.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Non Interventional — This is a non therapeutic, pilot study.

SUMMARY:
This is a non-interventional, R01-funded pilot study that will identify serum and cellular markers in patients' blood samples that can be used as short-term biomarkers of rituximab response. We hypothesize that serum complement levels, activation of natural killer cells, and clearance of peripheral B-cells will be accurate biomarkers of rituximab response, and may be correlated with long-term outcomes.

DETAILED DESCRIPTION:
This study does not involve the administration of study drug. This study will only require additional blood draws to identify how patients respond to rituximab and other anti-CD20 antibody therapy. It is expected that blood draws will occur on the same day in which an IV is placed to dose you with the anti-CD20 antibody or for other bloodwork being performed in order to avoid extra sticks.

If you take part in this study, you will have additional blood drawn at the following time-points surround anti-CD20 antibody therapy:

Pre Dose, Cycle 1

* Two 7.5 ml tubes (two teaspoons) of blood will be taken along with your other pre-chemotherapy bloodwork Post Dose, Cycle 1
* Two 5 ml tubes (three teaspoons) of blood will be taken Pre Dose, Cycle 2
* Two 5 ml tubes (two teaspoons) of blood will be taken Post Dose, Cycle 2
* Two 5 ml tubes (two teaspoons) of blood will be taken Pre Dose, Cycle 6
* Two 10 ml tubes (four teaspoons) of blood will be taken Post Dose, Cycle 6
* Two 10 ml tubes (four teaspoons) of blood will be taken

Note: Two tubes will be taken at each draw. If no blood was drawn in the prior 8 weeks, 10 ml of blood will be taken per tube. For the first 4 draws (at cycle 1 and cycle 2, pre- and post-), the amount of blood being taken is to ensure that the patient does not have more than 50 ml of blood taken within an 8 week period.

ELIGIBILITY:
Inclusion Criteria:

1. Any adult patient who has not received rituximab or other anti-CD20 antibody within the past year who is initiating rituximab or other anti-CD20 antibody treatment.
2. Treatment plan that includes at least two doses of anti-CD20 antibody and longitudinal follow up over at least a one-month time span.

Exclusion Criteria:

1. Hgb less than 8.0 g/dL or Hct less than 25% (transfusions or growth factors are permissible).
2. Treatment with any anti-CD20 antibody within the past 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any adult patient who has not received rituximab or other anti-CD20 antibody within the past year who is initiating rituximab or other anti-CD20 antibody treatment and has a treatment plan that includes at least two doses of anti-CD20 antibody and longitudinal follow up over at least a one-month time span.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2019-02-07 (Actual); Study Completion 2019-02-07 (Actual)

PRIMARY OUTCOMES:
Percentage of peripheral blood mononuclear cells that are B-cells, as measured by flow cytometry for CD19 performed on peripheral blood immediately prior to cycle 2 | 1 month after the start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ari M Melnick, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Medical College of Cornell University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No